CLINICAL TRIAL: NCT04844658
Title: A Comparative Randomized Clinical Study on Covid-19 Positive Hospitalized Patients Supplemented With NASAFYTOL
Brief Title: Covid-19, Hospitalized, PatIents, Nasafytol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilman S.A. (Industry)
Collaborators: Artialis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHOPIN
Record Dates: First submitted 2021-04-12; First posted 2021-04-14 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard treatment + NASAFYTOL® (Experimental): Minimum 25 patients will receive NASAFYTOL® as a supportive supplementation to standard treatment of hospitalized patients infected with COVID-19.
  For each patient, 8 capsules of NASAFYTOL® taken orally per day (4 capsules in the morning and 4 capsules in the evening before meal ,with a full glass of water. ) in support of the standard COVID-19 treatment in force in the hospital from the day after the randomization (day1) and during the period of hospitalization and maximum for 14 days
  Interventions: Dietary Supplement: NASAFYTOL®; Drug: Strandard of care treatment
- standard treatment + FULTIUM® - D3 800 (Active Comparator): Minimum 25 patients will receive vitamin D , FULTIUM® - D3 800 as a supportive supplementation to standard treatment of hospitalized patients infected with COVID-19.
  For each patient,1 capsule of Vitamin D taken orally per day (1 capsule in the morning) in support of the standard COVID-19 treatment in force in the hospital from the day after the randomization (day1) and for the duration of the hospitalization and maximum for 14 days
  Interventions: Dietary Supplement: FULTIUM® -D3 800; Drug: Strandard of care treatment

INTERVENTIONS:
Dietary Supplement: NASAFYTOL® — Dietary supplement presented as green soft gel capsules of 1008 mg, containing a bioactive mixture of turmeric extract or curcumin, natural quercetin from Sophora japonica L. and vitamin D3.
  Arms: standard treatment + NASAFYTOL®
Dietary Supplement: FULTIUM® -D3 800 — Vitamin D , FULTIUM® - D3 800 is a blue soft capsule that contains 800 UI (20 µg) of D3 vitamin (cholecalciferol).
  Arms: standard treatment + FULTIUM® - D3 800
Drug: Strandard of care treatment — Strandard of care treatment for Covid-19 infection

SUMMARY:
The objective of this study is to evaluate the effect and safety of NASAFYTOL® on COVID-19 positive hospitalized patients as a supportive supplementation to standard-of-care in improving clinical parameters safely during hospital admission (maximum 14 days).

The study is a standard-of-care comparative, open, parallel two-arms and randomized trial in 50 adult patients positive to COVID-19 infection and hospitalized. It will be monocentric but may be extended to several investigation sites (multicentric) depending on the evolution of the epidemic within the hospitals.

DETAILED DESCRIPTION:
50 patients (25 per arm) infected with COVID-19 and hospitalized (depending on the progress of the pandemic and therefore the presence of COVID-19 patients, this number could reach 100 (50 per arm)). The first ten sentinel patients will be monitored at the safety level before enrolling the rest of the participants.

The effect and safety of NASAFYTOL® will be evaluated using the following outcome measures:

1. Improvement of clinical condition of the patient defined by the COVID-19 WHO ordinal Outcomes score. This scale reflects a range from uninfected to dead, where 0 is "no clinical or virological evidence of infection", 1 is "no limitation of activities", 2 is "limitation of activities", 3 is "hospitalized, no oxygen therapy", 4 is "oxygen by mask or nasal prongs", 5 is "non-invasive ventilation or high-flow oxygen", 6 is "intubation and mechanical ventilation", 7 is "ventilation + additional organ support - pressors, RRT (renal replacement therapy), ECMO (extracorporeal membrane oxygenation)", and 8 is "death".

   * Time to a 1-point decrease
   * Score at 14 days (or at hospital leave if <14 days) post randomization
2. Duration (days) of hospitalization
3. In-hospital mortality
4. Temperature (fever):

   * Time to resolution of fever for at least 48 hours without antipyretics for 48 hours - Defined as ≤36.6°C (axilla), ≤37.2°C (oral) or ≤37.8°C (rectal or tympanic)
   * Proportion of participants with normalization at day 14 (or at hospital leave if <14 days)
5. Need of oxygen therapy
6. Tolerance as defined by the Incidence of Adverse Events (AE) and Serious Adverse Events (SAE)
7. Compliance using the pill count
8. Blood test:

   * C-reactive proteins : Time to halving of (or achieve normal ) CRP levels compared to peak value during trial
   * Hematological values (included Lymphocyte Count) and others routine laboratory parameters (LDH, albumin, etc.): Time to normalization
   * Vitamin D serum concentration: comparison of concentration between inclusion and end of trial and between the 2 arms.

   Optional outcome measures will be perform if data is available from routine practice:
9. Blood tests between inclusion and end of trial
10. Radiological response - Thoracic CT scan or Chest XR
11. Oxygenation PaO2 (partial pressure of oxygen) / FiO2 (fraction of inspired oxygen, FiO2) ratio (or P/F ratio) :

    * Time to improvement (TBD) in oxygenation for at least 48 hours
    * Proportion of participants with normalization at day 14 (or at hospital leave if <14 days)
12. Time until negative RT-PCR

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years of age at the time of inclusion in the study;
* Recently hospitalized patients in whom SARS CoV-2 infection has been laboratory confirmed by RT-PCR or other commercial or public health test on any sample.
* Severity of 3-4-5 according to the WHO 7-point ordinal scale (3: hospitalized, no oxygen therapy; 4: hospitalized, oxygen by mask or nasal prongs; 5:non-invasive ventilation or high-flow oxygen);
* Subject (or authorized legal representative) who can provide oral or written informed consent before beginning any study procedure;
* Understand and agree to abide by the study procedures.

Exclusion Criteria:

* Contra-indication to NASAFYTOL® or constituents (incl. Vit D): hypersensitivity or allergy to product components;
* Swallowing disorder or inability to take oral caps;
* Presence of comorbidities that imply a poor prognosis (according to clinical judgment);
* Pregnancy or breastfeeding women; If patient is a female of childbearing potential, patient must use an effective means of birth control (oral, intravaginal or transdermal oestrogen-progestogen combined hormonal contraceptives or intrauterine devices or sexual abstinence);
* Serious or active bacterial infections or documented sepsis by pathogens other than SARS-CoV-2;
* Patients participating in clinical trials of other products; Patients presenting acute impairment of renal function or nephrolithiasis; ALT/AST> 5 times the normal limit, or Neutropenia (Absolute neutrophil count < 500/uL), or Thrombocytopenia (Platelets < 50,000/uL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Improvement of the patient's clinical condition based on the WHO ordinal outcomes score | day 14
  Time to a 1-point decrease on the ordinal scale. The ordinal scale reflects a range score from uninfected to dead, where 0 is "no clinical or virological evidence of infection", 1 is "no limitation of activities", 2 is "limitation of activities", 3 is "hospitalized, no oxygen therapy", 4 is "oxygen by mask or nasal prongs", 5 is "non-invasive ventilation or high-flow oxygen", 6 is "intubation and mechanical ventilation", 7 is "ventilation + additional organ support - pressors, RRT (renal replacement therapy), ECMO (extracorporeal membrane oxygenation)", and 8 is "death".
Improvement of the patient's clinical condition based on the WHO ordinal outcomes score | day 14
  Ordinal score at 14 days (or at hospital leave if <14 days) post randomization. The ordinal scale reflects a range score from uninfected to dead, where 0 is "no clinical or virological evidence of infection", 1 is "no limitation of activities", 2 is "limitation of activities", 3 is "hospitalized, no oxygen therapy", 4 is "oxygen by mask or nasal prongs", 5 is "non-invasive ventilation or high-flow oxygen", 6 is "intubation and mechanical ventilation", 7 is "ventilation + additional organ support - pressors, RRT (renal replacement therapy), ECMO (extracorporeal membrane oxygenation)", and 8 is "death".
Duration of hospitalization | day 14
  Number of days hospitalization
In-hospital mortality | day 14
  Number of deads
Temperature (fever) | day 14
  Time to resolution of fever for at least 48 hours without antipyretics for 48 hours - Defined as ≤36.6°C (axilla), ≤37.2°C (oral) or ≤37.8°C (rectal or tympanic)
Temperature (fever) | day 14
  Proportion of participants with normalization at day 14 (or at hospital leave if <14 days)
Need of oxygen therapy | day 14
  Proportion of participants with oxygen therapy
Tolerance as defined by the Incidence of Adverse Events (AE) | day 14
  Numbers of Adverse Events
Tolerance as defined by the incident of Serious Adverse Events (SAE) | day 14
  Numbers of Serious Adverse Events
Compliance using the pill count | day 14
  Numbers of Pill count taken by the patient
Blood test | day 14
  C-reactive proteins : Time to halving of (or achieve normal ) CRP levels compared to peak value during trial
Blood test | day 14
  Hematological values (included Lymphocyte Count) and others routine laboratory parameters (LDH, albumin, etc.): Time to normalization
Blood test | day 14
  Vitamin D serum concentration: comparison of concentration between inclusion and end of trial and between the 2 arms.

OTHER OUTCOMES:
Radiological response (exploratory) | day 14
  Thoracic CT scan or Chest XR if available
Oxygenation | day 14
  Time to improvement in oxygenation ratio for at least 48 hours. PaO2 (partial pressure of oxygen) / FiO2 (fraction of inspired oxygen, FiO2) ratio (or P/F ratio)
Oxygenation | day 14
  Proportion of participants with ratio normalization at day 14 (or at hospital leave if <14 days) PaO2 (partial pressure of oxygen) / FiO2 (fraction of inspired oxygen, FiO2) ratio (or P/F ratio)

CONTACTS AND LOCATIONS:
Locations (1):
- Delta Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerain J, Uebelhoer M, Costes B, Herman J, Pietri S, Donneau AF, Monseur J, Henrotin Y. NASAFYTOL(R) supplementation in adults hospitalized with COVID-19 infection: results from an exploratory open-label randomized controlled trial. Front Nutr. 2023 Jun 22;10:1137407. doi: 10.3389/fnut.2023.1137407. eCollection 2023. PMID 37426178